CLINICAL TRIAL: NCT05480462
Title: Single Blind, Randomized, Comparative, Multicentre Clinical Trial of the Immunogenicity and Safety of Booster Immunization With Bivalent Vaccine Against Tetanus and Diphtheria CLODIVAC (IBSS Biomed S.A.) and Td-Impfstoff Mérieux (Sanofi Pasteur) in Healthy Adults.
Brief Title: Immunogenicity and Safety of Vaccine Against Tetanus and Diphtheria.
Acronym: Clodivac
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: IBSS Biomed S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21-BIO-0002
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Diphtheria; Tetanus
Keywords: Vaccine; Booster
MeSH Terms: conditions — Diphtheria; Tetanus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clodivac (Experimental)
  Interventions: Biological: Clodivac
- Td-Impfstoff Merieux (Active Comparator)
  Interventions: Biological: Td-Impfstoff Merieux

INTERVENTIONS:
Biological: Clodivac — A dose of 0.5 ml should be administered intramuscularly into deltoid muscle.
  Arms: Clodivac
Biological: Td-Impfstoff Merieux — One dose (0.5 ml) intramuscular, preferably in the deltoid muscle of the upper arm.
  Arms: Td-Impfstoff Merieux

SUMMARY:
A single blind, randomized, comparative, multicentre clinical trial of the immunogenicity and safety of booster immunization with bivalent vaccine against tetanus and diphtheria CLODIVAC (IBSS BIOMED S.A.) and Td-Impfstoff Mérieux (Sanofi Pasteur) in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Approved informed consent.
2. Men and women aged 18- 65 years.
3. Written confirmation on previous immunization against diphtheria and tetanus not older than 16 years and not younger than 4 years.

Exclusion Criteria:

1. Subject with acute infectious diseases.
2. Subject allergic to any of the substances of the IMP administered in clinical trial.
3. Subject with Guillain-Barré syndrome or neuropathy, an anaphylactic or other allergic reactions after previous vaccination against tetanus or diphtheria.
4. Subject with primary or secondary immunodeficiency (e.g. congenital immunodeficiency, HIV infection, organ or bone marrow transplantation, leukemia, lymphoma, Hodgkin's disease, multiple myeloma, generalized malignancy, drugs or other causes induced immunodeficiency).
5. Subject with progressive or unstable neurological disorder.
6. Subject with severe thrombocytopenia or any coagulation disorder not allowing the intramuscular administration.
7. Subject with blood product treatment, including immunoglobulins within the last 90 days prior to study entry.
8. Subject vaccinated less than 14 days inactivated or live vaccine prior to study entry.
9. Pregnant woman and breastfeeding (anamnestically).
10. Subject incapable of cooperation.
11. Alcohol or drug abuse.
12. Subject currently participating in another clinical trial or in drug evaluation, within 4 weeks prior to study entry.
13. Subjects requiring vaccination against tetanus after severe injury.
14. Any other condition that in the Investigator's opinion may affect the safety of the test participant or the integrity of data obtained during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-03-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Seroconversion | 28 days
  The primary endpoint is the seroconversion in 28 days follow-up. The proportion of subjects complying the positive criteria of seroconversion will be calculated.

SECONDARY OUTCOMES:
The ratio of geometric mean concentrations (GMC) of post-vaccination tetanus antibodies and diphtheria antibodies between test and reverence. | 28 days
  1. The ratio of geometric mean concentrations (GMC) of post-vaccination tetanus antibodies between test and reference vaccine in 28 days FU.
  2. The ratio of geometric mean concentrations (GMC) of post-vaccination diphtheria antibodies between test and reference va1. The ratio of geometric mean concentrations (GMC) of post-vaccination tetanus antibodies between test and reference vaccine in 28 days FU.

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - SPZOZ w Bochni Szpital Powiatowy im. bł. M. Wieckiej, Bochnia
  - Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow

IPD SHARING:
Plan to Share IPD: No